CLINICAL TRIAL: NCT06020781
Title: Efficacy and Safety of Dexmedetomidine to 20ml Bupivacaine in Supraclavicular Brachial Plexus Block
Brief Title: Efficacy and Safety of Dexmedetomidine to Bupivacaine in Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Gamal Hendawy Shams, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine Faculty of Medicine Kafr-El Sheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-51
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Dexmedetomidine; Bupivacaine; Supraclavicular Brachial Plexus Block
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine and Dexmedetomidine (Experimental): Patients will receive ultrasound-guided Supraclavicular brachial plexus block with 20 ml bupivacaine 0.5% + 1 μg/kg dexmedetomidine.
  Interventions: Drug: bupivacaine and dexmedetomidine.
- 20 ml Bupivacaine without additives (Active Comparator): Patients will receive ultrasound-guided Supraclavicular brachial plexus block with 20 ml bupivacaine 0.5% without additives.
  Interventions: Drug: bupivacaine only
- 30 ml bupivacaine without additives (Active Comparator): Patients will receive ultrasound-guided Supraclavicular brachial plexus block with 30 ml bupivacaine 0.5% without additives as a control group.
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: bupivacaine and dexmedetomidine. — patient will receive Ultrasound -guided Supraclavicular brachial plexus block with 20 ml bupivacaine 0.5% + 1 μg/kg dexmedetomidine.
  Arms: Bupivacaine and Dexmedetomidine
Drug: bupivacaine only — patient will receive Ultrasound -guided Supraclavicular brachial plexus block with 20 ml bupivacaine 0.5% without additives
  Arms: 20 ml Bupivacaine without additives
Drug: bupivacaine — patient will receive Ultrasound -guided Supraclavicular brachial plexus block with 30 ml bupivacaine 0.5% without additives as a control group.
  Arms: 30 ml bupivacaine without additives

SUMMARY:
The study aims to evaluate the analgesic efficacy and safety of addition of 1µg/kg dexmedetomidine to 20ml bupivacaine compared to 20ml and 30ml bupivacaine without additives in ultrasound-guided supraclavicular brachial plexus block for anesthesia.

DETAILED DESCRIPTION:
Dexmedetomidine, a highly selective α2 adrenergic agonist, has been used as an adjuvant to local anesthetics. Various clinical trials performed have shown dexmedetomidine to be safe when used as an adjuvant to local anesthetic in subarachnoid, caudal, and epidural Different doses of dexmedetomidine are commonly used as an additive in Ultrasound-guided supraclavicular brachial plexus block, 1 μg/kg and 2 μg/kg in which a high dose of dexmedetomidine does not prolong the duration of analgesia, but it is associated with lower heart rate and blood pressure. Incidence of hypotension and bradycardia is also more. Hence, a lower dose of 1 μg/kg dexmedetomidine is a good balance between safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) grade I or II patients
* both sexes
* scheduled for elective upper limb surgery below mid-humerus level under Ultrasound -guided Supraclavicular brachial plexus block .

Exclusion Criteria:

* with pre-existing peripheral neuropathy of upper limb.
* Bleeding disorders.
* Infection at injection site.
* Untreated pneumothorax.
* Patients on adrenoreceptor agonist or antagonist therapy.
* History of severe cardiac,.respiratory, hepatic, or renal disease.
* pregnancy and known hypersensitivity to the study drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Success rate. | 30 minutes after block performance
  Sensory and motor block evaluation will be done every 3 min after giving the block until complete sensory and motor block or 30 min, whichever will be earlier.

SECONDARY OUTCOMES:
Total pethidine consumption. | 24 hours postoperative.
  Visual analog scale ≥ 4 indicates the analgesic requirements. The patient will be given supplementary pethidine I.V. injection in a dose of 0.5 mg as rescue analgesia. Total pethidine consumption postoperative in the 1st 24 hours will be measured.
Pain score. | 24 hours postoperative.
  Pain score will be measured by visual analogue scale (VAS) at 30 minutes and then at 2, 4, 6, 12, 18 and 24 hours postoperative.
  The VAS consists of a 10cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be).
Mean arterial blood pressure | From preoperatively till the end of surgery
  Mean arterial blood pressure from preoperatively, after block, then every 15 minutes intraoperative till the end of surgery.
Heart rate | From preoperatively till the end of surgery
  Heart rate from preoperatively, after block, then every 15 minutes intraoperative till the end of surgery.
Postoperative side effects. | 24 hours postoperative
  Complication related to the block or adverse events of the administered drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.